CLINICAL TRIAL: NCT05139966
Title: Eficácia de dentifrício Com Sistema de liberação Controlada de flúor Para remineralização de lesões Iniciais de cárie: Estudo clínico Randomizado.
Brief Title: Fluoride Controlled-release System for Initial Lesions of Caries
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Fabio Correia Sampaio, Titular Professor of Cariology Clinic, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NaFnano brushing
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: White Spot Lesion
Keywords: fluorine; dental plaque; Toothbrushing
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: A randomized, triple-blind crossover clinical trial study was performed to evaluate the bioavailability of intraoral fluoride in biomarkers of exposure (biofilm and saliva) after the use of mouthwash with experimental fluoride for one week, with wash-out periods between them
Who Masked: Care Provider
Masking Description: The products have a serial number and different colors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- G0 - placebo (Placebo Comparator): All placebo mouthwashes were formulated with the following common ingredients: WATER (AQUA), POLYSORBATE 80, HYDROXYPROPYL GUAR,,SODIUM BENZOATE, POTASSIUM SORBATE. Finally, NO FLUORIDE WAS INCORPORATED.
  Interventions: Drug: Mouthwash Product
- G1: 100% - sodium fluoride (100% free NaF) (Experimental): These mouthwashes were formulated with the following common ingredients: WATER (AQUA), POLYSORBATE 80, HYDROXYPROPYL GUAR,,SODIUM BENZOATE, POTASSIUM SORBATE. Finally, 225 ppm NaF (SODIUM FLUORIDE) WAS INCORPORATED.
  Interventions: Drug: Mouthwash Product
- G2: 50% nano fluoride (225 ppm, 50% free NaF + 50% nanoF) (Experimental): These mouthwashes were formulated with the following common ingredients: WATER (AQUA), POLYSORBATE 80, HYDROXYPROPYL GUAR,,SODIUM BENZOATE, POTASSIUM SORBATE. Finally, 225 ppm (50% free NaF + 50% nanoF) WAS INCORPORATED.
  Interventions: Drug: Mouthwash Product
- G3: 100% nano fluoride (225 ppm) (Experimental): These mouthwashes were formulated with the following common ingredients: WATER (AQUA), POLYSORBATE 80, HYDROXYPROPYL GUAR,,SODIUM BENZOATE, POTASSIUM SORBATE. Finally, 225 ppm (100% nanoF) WAS INCORPORATED.
  Interventions: Drug: Mouthwash Product

INTERVENTIONS:
Drug: Mouthwash Product — The participants were requested to rinse 10 ml of the mouthwash 2 times / day (morning and evening) for 1 min after toothbrushing (a non-F dentifrice was used throughout the study).
  Other Names: nano fluoride

SUMMARY:
OBJECTIVE: To evaluate in vivo the efficacy of fluoride-containing dentifrice incorporated in a controlled-release system (F-CSL, patent pending) in the remineralization of white spot lesions of caries in caries-active individuals. METHODS: A double-blind randomized clinical trial to evaluate the bioavailability of intraoral fluoride in biomarkers of exposure (biofilm and saliva) after the use of experimental toothpaste in the control of dental caries. The study will last three months. The participants of the study will be divided into three groups according to the dentifrice used. The sample will be selected randomly and composed of children and adolescents who seek the service of cariology of the UFPB. There will be participants of both sexes, preferably of the metropolitan region of João Pessoa in order to guarantee the low fluorine exposure by the water of supply. Intrabucal photographs will be obtained. Samples of saliva will be collected after 3 hours of the last meal. The benefits will be achieved by obtaining the reduction of the white spot area (mm2) plus the fact that all the children will be examined and will receive information on the treatment needs and forwading for the same.

DETAILED DESCRIPTION:
Study Design:A randomized, triple-blind crossover clinical trial study was performed to evaluate the bioavailability of intraoral fluoride in biomarkers of exposure (biofilm and saliva) after the use of mouthwash with experimental fluoride for one week, with wash-out periods between them. The biofilm was collected 1 hour (h) and 12h after toothbrushing and the use of mouthwash, and saliva was collected 1h (T1 - T60 min) and 12h. The data was obtained by potentiometry (ion selective electrode) for fluoride in these samples. The pilot test was performed with three participants before the study begins.

Experimental mouthwashes:The participants were allocated randomly to use the following experimental mouthwashes: P - placebo (without F); 100% sodium fluoride (NaF) (225 ppm) - positive control; 50% nanoencapsulated fluoride (225 ppm, 50% free NaF + 50% nanoF); and 100% nanoF (225 ppm) (Savoy SA - São Paulo, Brazil). All mouthwashes were packed in similar containers and had the same color and flavor. They were coded by an independent investigator not involved in the trial.

A simple randomization was performed taking into account a cross design. The unit of randomization was "mouthwash", so all mouthwashes had the same chance of being selected. The design of the study was created for each participant and for each new one another draw was made.

Clinical stage:First, the participants were submitted to dental prophylaxis and scraping to remove all biofilm and dental calculus. They used a placebo mouthwash for 7 days. Then, the Whitford protocol was followed [17]. Briefly, the subjects were instructed to rinse 10 ml of the mouthwash 2 times / day (morning and evening) for 1 min after toothbrushing (a non-F dentifrice was used throughout the study). On the seventh day, the subjects were instructed to brush only the occlusal surfaces, rinse the mouthwash 2 times and do not use dental floss, to allow biofilm accumulation. After going to bed, they abstained from eating or drinking anything except water, did not brush their teeth or use the mouthwash. The next morning, after 12 hours of last brushing and mouthwash, and fasting, the first samples of stimulated saliva and biofilm (upper and lower right hemi-arch) were collected. Then, the volunteers brushed the occlusal surfaces and rinsed 10 mL of the mouthwash for 1 min. Soon after, saliva samples were collected in the following times: t1, t5, t10, t15, t20, t30, t45 and t60 minutes. Later, 1 hour after the mouthwash, the biofilm samples (left side) were collected.

The stimulated saliva (chewing on a silicone) was collected for 2 min, posteriorly the saliva samples were centrifuged at 6,000 rpm for 10 minutes in order to separate the saliva debris. The biofilm was collected from all tooth surfaces, in both buccal and lingual areas, using a 3S hollenback spatula, from which the samples were immediately transferred to an eppendorff tube, centrifuged, subsequently dried at 60 °C for 4 h and then weighed.

Determination of the concentration of fluoride:The samples were analyzed by the hexamethyldisiloxane (HMDS) facilitated diffusion method of Taves [21] modified by Whitford [22]. The analyzes were performed with a fluoride specific electrode (model 9409; Orion Research) and a potentiometer (model EA 940; Orion Research, Cambridge, MA, USA) (Model 720 A Orion). Fluoride standards (1-100 nM) were used to prepare calibration curves.

Statistical analysis:Statistical analysis were performed in software R considering α = 0.05. The Shapiro-Wilk and Kolmogorov Smirnov tests were applied to evaluate the normality of the data. The comparisons of F concentration in saliva and biofilm between groups were performed by repeated measures ANOVA after the Bonferroni test. The AUC measure (area below the curve) was calculated to indicate the efficacy of F retention in the saliva over the long term by taking the F concentration values in the time interval from 12h to 60 min after the last rinse. The relationship between fluoride concentrations in biofilm and saliva was determined using Spearman's correlation coefficient. The data was calculated on Graph Pad Prism (version 6) and Statistical Package (SPSS) version 23.

ELIGIBILITY:
Inclusion Criteria:

* residents of a city without water fluoridation program

Exclusion Criteria:

* The use of orthodontic appliances, smokers, treatment with fluoride products and / or the use of antimicrobial in the last 4 weeks, carious lesions, periodontal disease and dental sensitivity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
levels of fluoride concentration in saliva and biofilm | 12 hours
  It is expected that a concentration of fluoride would differ according to the type of formulation providing beneficial support in remineralization of the tooth enamel and preventing carious lesions.

CONTACTS AND LOCATIONS:
Overall Officials: FABIO C SAMPAIO, PhD, Principal Investigator — Hospital Universitário Lauro Wanderley
Locations (1):
- Federal University of Paraíba, João Pessoa, Paraíba, Brazil